### 16-003707

### Latinas LEarning About Density (LLEAD Study)

NCT02910986

Document Date: 07/18/2019



Fecha de aprobación: 18 de julio de 2019 Válido hasta: 17 de julio de 2020

# FORMULARIO DE CONSENTIMIENTO PARA PARTICIPAR EN UN ESTUDIO Y AUTORIZACIÓN DE PRIVACIDAD

Nombre del estudio: Estudio para mujeres latinas que aprenden sobre la densidad mamaria

(Estudio LLEAD o Latinas Learning about Density)

**IRB N.º:** 16-003707

Investigadora principal: Dra. Celine Vachon y colegas

Por favor lea atentamente esta información que le comunica asuntos importantes sobre el estudio. Un miembro del equipo del estudio conversará con usted respecto a su participación en el mismo. Si en algún momento tiene alguna pregunta, por favor consúltenos.

Tómese su tiempo para decidir y converse libremente sobre el estudio con familiares, amigos y el proveedor de atención médica, antes de tomar su decisión.

A fin de ayudarla a decidir si desea tomar parte en este estudio, usted necesita saber lo siguiente:

- Participar en este estudio es un acto completamente voluntario.
- Puede elegir no participar.
- Si elige participar, puede cambiar de opinión en cualquier momento.
- Su decisión no ocasionará ninguna penalidad ni la hará perder los beneficios a los que, por lo demás, tiene derecho.
- Si decide no participar o suspende su participación, esa decisión no alterará la posibilidad de recibir atención médica en Mayo Clinic ahora, ni en el futuro.

Para fines de este formulario, Mayo Clinic se refiere a Mayo Clinic en Arizona, Florida y Rochester (Minnesota), al Sistema de Salud de Mayo Clinic y a todos los hospitales, clínicas afiliadas, hospitales y entidades que le pertenecen.

Si decide tomar parte en el estudio, usted firmará este consentimiento como demostración de que desea participar. Se le entregará una copia de este formulario.

Si quien firma este formulario de consentimiento lo hace en nombre de otra persona, la palabra "usted" que se utiliza en el formulario de consentimiento se refiere al participante.

IRB: 16-003707 01 Página 1 de 10 IRB Doc. Ctrl N.º 10013.28



Fecha de aprobación: 18 de julio de 2019 Válido hasta: 17 de julio de 2020 Nombre y número clínico

#### **INFORMACIÓN DE CONTACTO**

| Puede contactar a: | Al: | Si tiene preguntas acerca de: |
|---|---|---|
| Investigador(es) | Teléfono: | <ul> <li>Análisis y procedimientos del</li> </ul> |
| principal(es): | 507-284-9977 | estudio |
| Dra. Celine Vachon | | <ul><li>Lesiones o emergencias</li></ul> |
| Mayo Clinic de Rochester | | relacionadas con la investigación • Cualquier inquietud o duda |
| Dr. Bhavika Patel | Teléfono: | relacionada con el estudio |
| Mayo Clinic de Arizona | 480-301-7629 | <ul> <li>Retirarse del estudio</li> </ul> |
| , | | <ul> <li>Materiales recibidos</li> </ul> |
| Contacto para el equipo del estudio: | | ■ Citas relacionadas con el estudio |
| Edna Ramos | Teléfono: | |
| Arizona | 480-342-6112 | |
| 1 11 12 0 11 10 | 100 0 12 0112 | |
| | Nombre y dirección de la | |
| | institución: | |
| | Mayo Clinic Rochester | |
| | 200 1 <sup>st</sup> St SW | |
| | Rochester, MN 55906 | |
| | Mayo Clinic Arizona | |
| | 5777 E Mayo Blvd | |
| | Mayo Clinic Building | |
| | Phoenix, AZ 85054 | |
| | Teléfono: | <ul> <li>Derechos del participante en un</li> </ul> |
| Junta de Revisión | 507-266-4000 | estudio |
| Institucional (IRB) de Mayo | | |
| Clinic | Llamada gratuita: | |
| | 866-273-4681 | |
| | Teléfono: | ■ Derechos del participante en un |
| | 507-266-9372 | estudio |
| Defensor de los sujetos en | | <ul> <li>Cualquier inquietud o queja</li> </ul> |
| estudios (que no pertenece | Llamada gratuita: | relacionada con el estudio |
| al equipo del estudio) | 866-273-4681 | <ul> <li>Uso de información médica</li> </ul> |
| | | confidencial |
| | | <ul> <li>Retirar la autorización para utiliza</li> </ul> |



Fecha de aprobación: 18 de julio de 2019 Válido hasta: 17 de julio de 2020

| Puede contactar a: | Al: | Si tiene preguntas acerca de: |
|---|---|---|
| | Correo electrónico: researchsubjectadvocate@mayo.edu | su información médica confidencial |
| Facturación del estudio | Rochester, MN: 507-266-5670 Arizona: 800-603-0558 Asuntos de facturación o d seguro de salud relacionad el estudio | |

#### Otra información:

Una descripción de este ensayo clínico estará disponible en <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, según lo requieren las leyes de Estados Unidos. Ese sitio web no incluirá información que pueda identificarla; sino que, a lo más, incluirá un resumen de los resultados. Usted puede buscar en ese sitio web siempre que desee.

#### 1. ¿Por qué se le solicita participar en este estudio?

Se le solicita participar en este estudio porque usted tiene entre 40 y 74 años de edad y se hace una detección por mamografía.

Pueden participar 2000 pacientes en este estudio realizado en colaboración por Mayo Clinic y el Centro de Salud de Mountain Park.

#### 2. ¿Por qué se realiza este estudio?

Los resultados de la mamografía ahora informan a las mujeres acerca de su densidad mamaria. El propósito de este estudio es examinar tres maneras diferentes de comunicar esa información. Este estudio permitirá determinar si una de ellas es mejor que las otras para ayudar a que las mujeres entiendan sus resultados sobre la densidad mamaria y cuánto cuesta brindar esa información. Este estudio contribuirá nueva información respecto a la forma como las mujeres entienden la densidad mamaria y ayudará a determinar la mejor manera de brindar esa información a las pacientes. Además, se usará la información recolectada en el estudio para abordar otras preguntas acerca de la densidad mamaria, entre ellas, cuál es su relación con otros factores del estilo de vida y de riesgo clínico para cáncer de mama.

IRB: 16-003707 01 Página 3 de 10 IRB Doc. Ctrl N.º 10013.28



Fecha de aprobación: 18 de julio de 2019 Válido hasta: 17 de julio de 2020 Nombre y número clínico

#### 3. Información que usted debe conocer

#### ¿Quién financia el estudio?

Un subsidio de los Institutos Nacionales de Salud financiará este estudio.

#### 4. ¿Cuánto tiempo estará usted en el estudio?

Se le solicitará que participe en este estudio durante 5 años, a partir de la fecha en que reciba la notificación sobre su densidad mamaria.

#### 5. ¿Qué ocurrirá con usted durante su participación en el estudio?

Si usted califica para este estudio, se le solicitará que llene tres encuestas. La primera encuesta se hará en cuanto usted se inscriba en el estudio y le tomará aproximadamente 20 minutos llenarla.

La segunda encuesta se hará después de que usted reciba los resultados de la mamografía, o sea aproximadamente 2 semanas después de la mamografía. La coordinadora clínica del estudio (CRC, por sus siglas en inglés) se comunicará con usted por teléfono o correo para que llene la encuesta.

La tercera y última encuesta se llevará a cabo aproximadamente 1 año después de que usted reciba los resultados de la mamografía. La coordinadora clínica del estudio se comunicará con usted por teléfono o correo y le hará preguntas acerca de cómo se siente por los resultados y cuáles son sus planes para hacerse una mamografía u otros exámenes adicionales de detección del cáncer de mama en el futuro.

Podemos revisar su expediente médico para estudiarlo. Podemos también solicitarle autorización para recolectar sus expedientes médicos de otros proveedores de atención médica y revisarlos. Solamente recolectaremos y revisaremos los expedientes correspondientes a los exámenes o análisis para detección del cáncer de mama relacionados con las citas de seguimiento para la salud de las mamas y la densidad mamaria.



| Nombre y número clínico |
|-------------------------|

Fecha de aprobación: 18 de julio de 2019 Válido hasta: 17 de julio de 2020

Como parte de su atención clínica habitual, se le hará una mamografía normal y los resultados los recibirá igual, sea que decida participar o no en el estudio. Si decide participar en este estudio, recibirá más información educativa por escrito junto con los resultados de la mamografía, o una *promotora* (educadora sobre la salud bilingüe) puede comunicarse con usted por teléfono para hablar sobre los resultados de la mamografía, además de recibirlos. Estamos estudiando 3 maneras diferentes de entregar los resultados sobre la densidad mamaria a las pacientes y, por ello, se asignará a las mujeres que participan en este estudio a una de las tres maneras de recibir los resultados de la mamografía. La determinación de que usted reciba más información educativa acerca de la densidad mamaria o de que se la llame por teléfono con los resultados de la mamografía será aleatoria (al azar):

- Usted tiene 1 probabilidad en 3 de recibir los resultados de la mamografía como normalmente lo hace, sin ninguna otra información educativa por escrito.
- Usted tiene 1 probabilidad en 3 de recibir los resultados de la mamografía junto con más información educativa escrita acerca de la densidad mamaria.
- Usted tiene 1 probabilidad en 3 de recibir los resultados de la mamografía junto con más información educativa escrita acerca de la densidad mamaria y una llamada de la *promotora* para hablar sobre la información.

En las mujeres del tercer grupo, algunas de las llamadas telefónicas con la *promotora* se grabarán con el fin de garantizar la calidad. Esas llamadas también se revisarán para fines del estudio, por ejemplo, para entender mejor las preguntas femeninas acerca de la densidad mamaria. En caso de que se la asigne al tercer grupo, que incluye la llamada de la *promotora*, por favor seleccione su respuesta a continuación:

Estoy dispuesta a permitir que mi conversación telefónica con la *promotora* sea grabada:

| Por favor marque una casilla: | | | |
|---|---|---|---|
| | ☐ Sí | No Escriba sus iniciales aquí: | Fecha: |
| 6. | ¿Cuáles so<br>estudio? | n los posibles riesgos o molest | tias de su participación en el |

El presente estudio es de riesgo mínimo. No conlleva ningún riesgo de importancia el hecho de llenar las encuestas ni de revisar los expedientes médicos. Es posible que algunas de las preguntas de las encuestas acerca de cómo se siente usted o qué está pensando puedan parecerle muy personales, pero puede dejar sin respuesta cualquier pregunta que no desee responder.

IRB: 16-003707 01 Página 5 de 10 IRB Doc. Ctrl N.º 10013.28



Fecha de aprobación: 18 de julio de 2019 Válido hasta: 17 de julio de 2020

Las encuestas del estudio no formarán parte de su expediente médico y solo el personal del estudio tiene acceso a ellas. Toda la información y datos del estudio se guardarán en la base de datos sobre estudios que Mayo Clinic mantiene y que está protegida por una contraseña.

#### 7. ¿Existe alguna razón por la que usted podría retirarse antes del estudio?

Participar en este estudio es decisión suya. Usted puede decidir suspender su participación en cualquier momento.

#### 8. ¿Qué ocurre si usted sufre alguna lesión por participar en el estudio?

#### ¿Dónde puede recibir ayuda?

Si usted cree que sufrió alguna lesión relacionada con su participación en el estudio, debe notificarlo oportunamente a los investigadores principales, cuyos nombres aparecen bajo las personas de contacto al principio de este formulario. Mayo Clinic le ofrecerá atención médica para las lesiones relacionadas con el estudio, incluso primeros auxilios, tratamiento de emergencia y cuidados de seguimiento, según sea necesario.

¿Quién pagará por el tratamiento de las lesiones relacionadas con la investigación? Mayo brindará servicios médicos para el tratamiento de cualquier efecto secundario por la participación en el estudio. Dichos servicios serán gratuitos, si no están cubiertos por un plan de salud o seguro médico No se ofrecerá ningún otro dinero.

#### 9. ¿Cuáles son las posibles ventajas de participar en este estudio?

El presente estudio no mejorará su salud, pero tal vez la ayude a entender los resultados de la mamografía.

#### 10. ¿Qué otras alternativas tengo si opto por no participar en este estudio?

El estudio se realiza para recolectar información. Usted puede elegir no participar en el estudio.

IRB: 16-003707 01 Página 6 de 10 IRB Doc. Ctrl N.º 10013.28



Fecha de aprobación: 18 de julio de 2019 Válido hasta: 17 de julio de 2020

## 11. ¿Por cuáles análisis o procedimientos deberá usted pagar si participa en este estudio?

Usted deberá pagar por todos los exámenes y procedimientos que usted normalmente se haría como parte de su atención médica normal, incluida la mamografía.

#### 12. ¿Recibirá usted pago por su participación en este estudio?

Usted puede recibir una compensación máxima de 75 dólares al terminar el estudio.

Usted recibirá 25 dólares al terminar la primera encuesta; 25 dólares al terminar la segunda encuesta, aproximadamente 4 semanas después; y 25 dólares al terminar la tercera encuesta, aproximadamente un año después de recibir los resultados de la mamografía.

#### 13. ¿Cómo se protegerá la confidencialidad y privacidad de sus expedientes?

Mayo Clinic se compromete a proteger la confidencialidad de la información obtenida sobre usted relacionada con este estudio.

Las respuestas a las preguntas de las encuestas recibirán un código que se conectará con la información en una base de datos segura a la que solamente el personal del estudio puede acceder.

Durante el presente estudio, se recolectará información sobre su salud. Según la ley federal conocida como Regulación de Privacidad, la información de salud es confidencial; sin embargo, hay excepciones a esta regulación y usted necesita sabe quién puede ver, usar y compartir su información de salud para el estudio y por qué tendrían que hacerlo. La información sobre usted y su salud no puede usarse en este estudio sin su autorización escrita. Su firma en este formulario significa que usted otorga ese permiso.



Fecha de aprobación: 18 de julio de 2019 Válido hasta: 17 de julio de 2020

#### Se puede obtener información de salud suya de lo siguiente:

- Expedientes médicos anteriores, actuales y futuros.
- Procedimientos del estudio, lo que incluye visitas médicas, análisis, entrevistas y cuestionarios.

#### ¿Por qué se utilizará y/o entregará esta información a otros?

- A fin de realizar el estudio.
- A fin de informar sobre los resultados.
- A fin de ver si el estudio se realizó correctamente.

Si los resultados del estudio se hiciesen públicos, no se utilizará información que la identifique.

#### ¿Quién puede usar o compartir su información de salud?

- El personal de Mayo Clinic que participa en el presente estudio.
- Al firmar este formulario, usted brinda su permiso expreso al Centro de Salud de Mountain Park para que ofrezca a Mayo Clinic la información sobre su salud relacionada con este estudio.

#### ¿Con quién se podría compartir su información de salud?

- La Junta de Revisión Institucional de Mayo Clinic que supervisa el estudio.
- Los investigadores de otras instituciones que están involucrados en el estudio.
- Las agencias federales y estatales (tales como la Administración de Alimentos y Medicamentos, el Departamento de Salud y Servicios Humanos, los Institutos Nacionales de Salud y otras entidades estadounidenses), así como organizaciones gubernamentales de otros países que supervisan o revisan los estudios.
- El patrocinador o los patrocinadores del estudio y las personas o grupos que ellos contraten para ayudarles a llevar a cabo el estudio.
- Un grupo que supervisa los datos (información del estudio) y la seguridad de esta investigación.

## ¿Estará su información de salud protegida después de haberla compartido con otros?

Mayo Clinic solicita a todos los que reciben su información de salud que protejan su privacidad, pero una vez que se comparte la información fuera de Mayo Clinic, ya no es posible prometer que ésta permanecerá confidencial y existe la posibilidad de que para entonces tampoco esté protegida por la Regulación de Privacidad.

#### Sus derechos de privacidad

Usted no tiene obligación de firmar este formulario, pero si no lo hace, no podrá participar en el estudio.

IRB: 16-003707 01 Página 8 de 10 IRB Doc. Ctrl N.º 10013.28



Fecha de aprobación: 18 de julio de 2019 Válido hasta: 17 de julio de 2020

Si usted retira su autorización para usar o compartir la información sobre su salud, entonces concluirá su participación en este estudio y no se obtendrá más información suya, pero se continuará utilizando la información ya obtenida sobre usted.

Si decide no participar o retirarse del estudio, eso no repercutirá negativamente sobre la relación que usted mantiene con sus médicos ni con Mayo Clinic.

Usted puede revocar su autorización para usar o compartir información sobre su salud en cualquier momento, mediante el envío de una carta a la siguiente dirección:

Mayo Clinic Office for Human Research Protection ATTN: Notice of Revocation of Authorization 200 1st Street SW Rochester, MN 55905

De lo contrario, puede también revocar su autorización enviando un correo electrónico al defensor de los sujetos en investigaciones de Mayo Clinic, a: researchsubjectadvocate@mayo.edu.

Por favor verifique que su carta o correo electrónico contenga la siguiente información:

- El nombre del investigador principal.
- El número de IRB del estudio y/o el nombre del estudio.
- La información para entrar en contacto con usted.

Su autorización durará hasta el fin del estudio, a menos que usted la revoque. Debido a que el estudio es un proceso continuo, no es posible darle una fecha exacta para la finalización del estudio.



Fecha de aprobación: 18 de julio de 2019 Válido hasta: 17 de julio de 2020

| FIRMAS PARA LA INSCRIPCIÓN Y AUTORIZACIÓN: | | |
|---|---|---|
| Su firma documenta su autorización para participar en este studio. | | |
| Nombre en letra de imprenta | Fecha (mes,dia, año completo) | Hora (hh:mm, am/pm) |
| Firma | | |
| <ul> <li>Persona que obtiene el consenti</li> <li>Expliqué a la participante</li> <li>Respondí todas las pregur</li> </ul> | | o de mis capacidades. |
| Nombre en letra de imprenta | Fecha (mes, dia, año completo) | Hora (hh:mm, am/pm) |
| Firma | | |